CLINICAL TRIAL: NCT01707719
Title: Isolated Erythrocyte Membrane Susceptibility to Photo-oxidative Stress in Patients Affected by Alzheimer's Disease and Healthy Controls
Brief Title: Isolated Erythrocyte Membrane Susceptibility to Photo-oxidative Stress in Alzheimer's Disease
Status: Completed | Type: Observational
Sponsor: Raffaele Antonelli Incalzi (Other)
Responsible Party: Sponsor-Investigator, Raffaele Antonelli Incalzi, Professor, Campus Bio-Medico University
Organization: Campus Bio-Medico University (Other)
Other Study IDs: ERASE
Record Dates: First submitted 2012-10-01; First posted 2012-10-16 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2018-03

CONDITIONS: Alzheimer Disease; Oxidative Stress; Adrenocortical Hyperfunction
Keywords: Alzheimer's disease; Oxidative stress; HPA axis
MeSH Terms: conditions — Alzheimer Disease; Adrenocortical Hyperfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Alzheimer's disease
- Non demented subjects

SUMMARY:
High lipid peroxidation and altered antioxidant defenses have been frequently reported in Alzheimer's disease patients.

The purpose of this study is to investigate susceptibility to photo-oxidation of isolated erythrocyte membranes, in patients affected by Alzheimer's disease and age- and sex-matched, non demented subjects.

DETAILED DESCRIPTION:
The study hypothesis is that high lipid peroxidation and decreased antioxidant defenses characterize the natural history of Alzheimer's disease.

It will be evaluated the release of malondialdehyde (MDA) from ex-vivo photo-oxidized erythrocyte ghosts, through a very easy and convenient lab procedure for the preparation of erythrocyte membrane samples.

Isolated and purified red blood cell membranes will be in vitro exposed to oxidative stress by UV-B radiation. The extent of cell membrane damage will be quantified by the fluorometric determination of MDA.

Induction of oxidative stress through ultraviolet rays, unlike that obtained by chemical oxidizing agents, is fully controllable, since it produces effects only during irradiation. Moreover, using isolated erythrocyte membranes allows for a greater specificity in the evaluation of MDA produced, and reduces the amount of blood required for the assay.

A portion of the blood sample (500 µL) will be sent to the laboratory of Lipinutragen (spin-off of CNR- National Research Center Bologna, Italy) where an erythrocyte membrane lipidomic analysis will be performed for the characterization of membrane phospholipids, in order to determinate the different lipid components (saturated fatty acids, monounsaturated and polyunsaturated, trans fatty acids), each one characterized by a different oxidative reactivity.

Recently published papers showed a striking association between urinary excretion of cortisol and the increase of some markers of oxidative damage of DNA and RNA (in humans). This finding provides further support to the idea that chronic psychological stress, who is associated to hypercortisolemia, can lead to an acceleration of the aging process.

The brain is a major target of the effects of glucocorticoids (CCS). The harmful consequences of cortisol on the hippocampus (one of the first brain areas affected by Alzheimer's disease) are well known. Some studies showed inverse correlations between cortisol levels and neuropsychological performance in patients with depression, dementia as well as in people treated chronically with CCS.

Alzheimer's disease is associated with states of hypercortisolism. Nonetheless, so far, its correlation with the level of oxidative stress has not been studied. We will investigate the relationship between 24h excretion of urinary cortisol and the level of malondialdehyde, produced by isolated and purified red blood cell membranes, in vitro exposed to oxidative stress by UV-B radiation.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients of both sexes diagnosed with Alzheimer's disease according to NINCDS-ADRDA criteria.
* Age and sex-matched elderly subjects without dementia.

Exclusion Criteria:

* Recent neoplasia (< 1 year)
* Vitamin B12 deficiency, positive serology for syphilis, thyroid function abnormalities considered to be significant by the care provider.
* Use of vitamin or mineral supplements.
* Diagnosis of malnutrition (based on body mass index and total protein levels)
* Metabolic syndrome or diabetes.
* Hormonal replacement therapy.
* Smoking
* Chronic inflammatory disease (e.g. rheumatoid arthritis) and any other acute illness.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients meeting NINCDS-ADRDA criteria for Alzheimer's disease and age- / sex-matched elderly subjects without dementia, will be recruited from those referring neurologists or geriatricians on an outpatient basis
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2015-06; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Malondialdehyde assay | At the time of recruitment
  Isolated and purified red blood cell membranes will be in vitro exposed to oxidative stress by UV-B radiation. The extent of cell membrane damage will be quantified by the fluorometric determination of malondialdehyde.

SECONDARY OUTCOMES:
Relationship between urinary excretion of cortisol and levels of malondialdehyde | At the time of recruitment
  Hyperactivity of the hypothalamic pituitary adrenal axis has been frequently described in Alzheimer's disease. Recently published work reported an association between high secretion of cortisol and oxidative stress. We will investigate the relationship between 24 h excretion of urinary cortisol and the level of malondialdehyde, produced by isolated and purified red blood cell membranes, in vitro exposed to oxidative stress by UV-B radiation.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Maria Serino, M.D. PhD, Principal Investigator — Doctors in Italy; Chiara Fanali, PhD, Principal Investigator — University Campus Bio-Medico; Laura Dugo, PhD, Principal Investigator — University Campus Bio-Medico; Simone Grasso, PhD, Principal Investigator — University Campus Bio-Medico; Ettore Bergamini, M.D., Study Chair — University of Pisa; Francesca Ursini, M.D., Principal Investigator — University Campus Bio-Medico; Fabrizio Vernieri, M.D., Principal Investigator — University Campus Bio-Medico; Marina Dachà, BS.Pharm, Study Director — University Campus Bio-Medico; Silvia Bernardini, M.D., Principal Investigator — University Campus Bio-Medico; Valentina Pasqualetti, PhD, Principal Investigator — University Campus Bio-Medico
Locations (1):
- Policlinico Universitario Campus Bio-Medico, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mangialasche F, Polidori MC, Monastero R, Ercolani S, Camarda C, Cecchetti R, Mecocci P. Biomarkers of oxidative and nitrosative damage in Alzheimer's disease and mild cognitive impairment. Ageing Res Rev. 2009 Oct;8(4):285-305. doi: 10.1016/j.arr.2009.04.002. Epub 2009 Apr 17. PMID 19376275
- [Background] Markesbery WR. Oxidative stress hypothesis in Alzheimer's disease. Free Radic Biol Med. 1997;23(1):134-47. doi: 10.1016/s0891-5849(96)00629-6. PMID 9165306
- [Background] Perry G, Nunomura A, Hirai K, Zhu X, Perez M, Avila J, Castellani RJ, Atwood CS, Aliev G, Sayre LM, Takeda A, Smith MA. Is oxidative damage the fundamental pathogenic mechanism of Alzheimer's and other neurodegenerative diseases? Free Radic Biol Med. 2002 Dec 1;33(11):1475-9. doi: 10.1016/s0891-5849(02)01113-9. PMID 12446204
- [Background] Mecocci P. Oxidative stress in mild cognitive impairment and Alzheimer disease: a continuum. J Alzheimers Dis. 2004 Apr;6(2):159-63. doi: 10.3233/jad-2004-6207. PMID 15096699
- [Background] Polidori MC, Mecocci P. Plasma susceptibility to free radical-induced antioxidant consumption and lipid peroxidation is increased in very old subjects with Alzheimer disease. J Alzheimers Dis. 2002 Dec;4(6):517-22. doi: 10.3233/jad-2002-4608. PMID 12629261
- [Background] Galbusera C, Facheris M, Magni F, Galimberti G, Sala G, Tremolada L, Isella V, Guerini FR, Appollonio I, Galli-Kienle M, Ferrarese C. Increased susceptibility to plasma lipid peroxidation in Alzheimer disease patients. Curr Alzheimer Res. 2004 May;1(2):103-9. doi: 10.2174/1567205043332171. PMID 15975074
- [Background] Casado A, Encarnacion Lopez-Fernandez M, Concepcion Casado M, de La Torre R. Lipid peroxidation and antioxidant enzyme activities in vascular and Alzheimer dementias. Neurochem Res. 2008 Mar;33(3):450-8. doi: 10.1007/s11064-007-9453-3. Epub 2007 Aug 25. PMID 17721818
- [Background] Serra JA, Dominguez RO, de Lustig ES, Guareschi EM, Famulari AL, Bartolome EL, Marschoff ER. Parkinson's disease is associated with oxidative stress: comparison of peripheral antioxidant profiles in living Parkinson's, Alzheimer's and vascular dementia patients. J Neural Transm (Vienna). 2001;108(10):1135-48. doi: 10.1007/s007020170003. PMID 11725816
- [Background] Kawamoto EM, Munhoz CD, Glezer I, Bahia VS, Caramelli P, Nitrini R, Gorjao R, Curi R, Scavone C, Marcourakis T. Oxidative state in platelets and erythrocytes in aging and Alzheimer's disease. Neurobiol Aging. 2005 Jun;26(6):857-64. doi: 10.1016/j.neurobiolaging.2004.08.011. PMID 15718044
- [Background] Bermejo P, Gomez-Serranillos P, Santos J, Pastor E, Gil P, Martin-Aragon S. Determination of malonaldehyde in Alzheimer's disease: a comparative study of high-performance liquid chromatography and thiobarbituric acid test. Gerontology. 1997;43(4):218-22. doi: 10.1159/000213853. PMID 9222750
- [Background] Baldeiras I, Santana I, Proenca MT, Garrucho MH, Pascoal R, Rodrigues A, Duro D, Oliveira CR. Peripheral oxidative damage in mild cognitive impairment and mild Alzheimer's disease. J Alzheimers Dis. 2008 Sep;15(1):117-28. doi: 10.3233/jad-2008-15110. PMID 18780972
- [Background] Torres LL, Quaglio NB, de Souza GT, Garcia RT, Dati LM, Moreira WL, Loureiro AP, de Souza-Talarico JN, Smid J, Porto CS, Bottino CM, Nitrini R, Barros SB, Camarini R, Marcourakis T. Peripheral oxidative stress biomarkers in mild cognitive impairment and Alzheimer's disease. J Alzheimers Dis. 2011;26(1):59-68. doi: 10.3233/JAD-2011-110284. PMID 21593563
- [Background] Onaran I, Yalcin AS, Sultuybek G. Effect of donor age on the susceptibility of erythrocytes and erythrocyte membranes to cumene hydroperoxide-induced oxidative stress. Mech Ageing Dev. 1997 Nov;98(2):127-38. doi: 10.1016/s0047-6374(97)00078-x. PMID 9379709
- [Background] Garcia-Arumi E, Andreu AL, Lopez-Hellin J, Schwartz S. Effect of oxidative stress on lymphocytes from elderly subjects. Clin Sci (Lond). 1998 Apr;94(4):447-52. doi: 10.1042/cs0940447. PMID 9640351
- [Background] Davis KL, Davis BM, Greenwald BS, Mohs RC, Mathe AA, Johns CA, Horvath TB. Cortisol and Alzheimer's disease, I: Basal studies. Am J Psychiatry. 1986 Mar;143(3):300-5. doi: 10.1176/ajp.143.3.300. PMID 3953862
- [Background] Costantini D, Marasco V, Moller AP. A meta-analysis of glucocorticoids as modulators of oxidative stress in vertebrates. J Comp Physiol B. 2011 May;181(4):447-56. doi: 10.1007/s00360-011-0566-2. Epub 2011 Mar 18. PMID 21416253
- [Background] Joergensen A, Broedbaek K, Weimann A, Semba RD, Ferrucci L, Joergensen MB, Poulsen HE. Association between urinary excretion of cortisol and markers of oxidatively damaged DNA and RNA in humans. PLoS One. 2011;6(6):e20795. doi: 10.1371/journal.pone.0020795. Epub 2011 Jun 7. PMID 21687734